CLINICAL TRIAL: NCT04390269
Title: Various Molecular Markers With Predictive and Prognostic Significance in COVID-19 Outcome
Brief Title: Immunogenetics Predictors With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Elbendary, Professor of Tropical Medicine and Hepatogastroenterology, Mansoura University
Other Study IDs: R.20.05.830.R1
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-05

CONDITIONS: Genetic Predisposition to Disease
Keywords: COVID-19; CYTOKINES; CHEMOKINES; GENETIC POLYMORPHISM; Immunity
MeSH Terms: conditions — Genetic Predisposition to Disease; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biological sample will take for the following analysis
  1. Routine diagnostic analysis Routine Laboratory testing includes complete blood picture (CBC), C-reactive protein (CRP), liver function tests, Blood sugar, serum creatinine
  2. Routine molecular diagnostic analysis Routine molecular Laboratory testing includes Real-time PCR Detection for SARS-COV 2
  3. Laboratory investigation for candidate gene i. Nucleic Acid Extraction from peripheral blood: the first step will include High-quality total nucleic acid extraction covering DNA, RNA, non-coding RNA, and Micro RNA ii. Allelic discrimination using ABI 7500 real-time PCR. The host DNA will be genotyped for candidate genes using TaqMan® SNP genotyping assays
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infected group: The infected group will be classified according to the severity whether mild ,moderate or severe
- susceptible (non infected: This group either exposed and not infected .
- control group: normal control subject

SUMMARY:
Background: There is a current worldwide outbreak of the novel coronavirus Covid-19 which originated from Wuhan in China and has now spread to 6 continents including 210 countries. There is still a lack of any report about severe acute respiratory syndromes (SARS-CoV-2) genetic polymorphisms which are associated with the susceptibility to infection. In addition, gene polymorphisms of MBL (mannose-binding lectin) associated with antigen presentation are related to the risk of SARS-CoV infection. Aim: To investigate the association of different genetic markers of different mechanisms of viral pathogenesis with the outcome of COVID-19. Methods: The study will include one hundred patients diagnosed as COVID-19. Biological blood samples will be taken for routine diagnostic analysis, routine molecular testing using Real-time polymerase chain reaction (PCR), Allelic discrimination and genotyping analysis. Outcome: Different genetic markers could play a role in the outcome and prognosis of COVID-19 viral infection.

DETAILED DESCRIPTION:
There is a current worldwide outbreak of the novel coronavirus Covid-19 (coronavirus disease 2019; the pathogen called SARS-CoV-2; previously 2019-nCoV), which originated from Wuhan in China and has now spread to 6 continents including 210 countries. Coronaviruses (CoVs), is a large family of single-stranded RNA viruses, can infect animals and humans, causing respiratory, gastrointestinal, hepatic, and neurologic diseases. Coronaviruses are a group of enveloped viruses with a positive-sense single-stranded RNA genome (26-39 kb). Four coronavirus genera (α, β, γ, δ) have been determined so far, with human coronaviruses (HCoVs) detected in the α coronavirus (HCoV-229E and NL63) and β coronavirus (e.g MERS-CoV and SARS-CoV) genera. This isolated novel β-CoV shows less than 80% similarity to the sequence of two bat-derived severe acute respiratory syndromes (SARS)-like coronaviruses, bat-SL-CoVZC45 and bat-SL-CoVZXC21, and about 50% identity to the sequence of a middle east respiratory syndrome (MERS-CoV). Patients with COVID-19 show general clinical manifestations including fever, dry cough, dyspnea, myalgia, fatigue, normal or decreased leukocyte counts, and radiographic evidence of pneumonia. After the virus enters the host cells, the viral RNA genome is released into the cytoplasm and is translated into two polyproteins and structural proteins, after which the viral genome begins to replicate. When the virus enters the host cells, its antigen will be presented to the antigen presentation cells(APC), which is a central part of the body's anti-viral immunity. Antigenic peptides are presented by major histocompatibility complex (MHC; or human leukocyte antigen (HLA) in humans) and then recognized by virus-specific cytotoxic T lymphocytes (CTLs). Hence, the understanding of the antigen presentation of SARS-CoV-2 will help our comprehension of COVID-19 pathogenesis. However, there is still a lack of any report about SARS-CoV-2, we can get a lot of information from previous researches on SARS-CoV and MERS-CoV. The antigen presentation of SARS-CoV mainly depends on MHC I molecules, but MHC II also contributes to its presentation.

These findings may provide valuable information for the rational design of vaccines against SARS-CoV-2. One of the main mechanisms for ARDS is the cytokine storm, the deadly uncontrolled systemic inflammatory response resulting from the release of huge amounts of pro-inflammatory cytokines and chemokines by immune effector cells in SARS-CoV infection. Better survive in host cells, SARS-CoV and MERS-CoV use multiple strategies to avoid immune responses. The evolutionarily conserved microbial structures called pathogen-associated molecular patterns can be recognized by pattern recognition receptors (PRR).

The antigen presentation can also be affected by the coronavirus. For example, gene expression related to antigen presentation is down-regulated after MERS-CoV infection. Therefore, destroying the immune evasion of SARS-CoV-2 is imperative in its treatment and specific drug development.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (> 18 years old) with COVID 19 infection.The patients will be classified on the basis of the severity of the disease.

Exclusion Criteria:

* -patients have symptoms of fever and /or respiratory with negative PCR for COVID-19.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: They will evaluate the clinical usefulness of the application of different diagnostic tests, monitoring tools and therapeutic options in clinical practice to improve the disease outcomes and reduce the costs of the disease burdens.
  In brief, the approach will consist of the following steps:
  1. Early diagnosis of patients at risk of COVID 19 evolution and their surveillance and monitoring by different means.
  2. Specific laboratory analysis for different genetic molecular tests for COVID 19 infection.
  3. Monitoring the genetic molecular tests in the follow-up periods.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2022-05-09 (Estimated)

PRIMARY OUTCOMES:
for the patients | 2 years
  To assess genetic mutation via detection of genetic polymorphisms of ACE2 in patients and control to detect what alleles will be associated with the susceptibility to COVID-19 and what alleles will be associated with clearance or protection from infections. using allelic discrimination SSCP (i.e Real-time PCR and genetic sequencer).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud El-Bendary, M.D, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Zhang J, Zhou L, Yang Y, Peng W, Wang W, Chen X. Therapeutic and triage strategies for 2019 novel coronavirus disease in fever clinics. Lancet Respir Med. 2020 Mar;8(3):e11-e12. doi: 10.1016/S2213-2600(20)30071-0. Epub 2020 Feb 13. No abstract available. PMID 32061335
- [Background] Xu Z, Li S, Tian S, Li H, Kong LQ. Full spectrum of COVID-19 severity still being depicted. Lancet. 2020 Mar 21;395(10228):947-948. doi: 10.1016/S0140-6736(20)30308-1. Epub 2020 Feb 14. No abstract available. PMID 32066525
- [Background] Zheng HY, Zhang M, Yang CX, Zhang N, Wang XC, Yang XP, Dong XQ, Zheng YT. Elevated exhaustion levels and reduced functional diversity of T cells in peripheral blood may predict severe progression in COVID-19 patients. Cell Mol Immunol. 2020 May;17(5):541-543. doi: 10.1038/s41423-020-0401-3. Epub 2020 Mar 17. No abstract available. PMID 32203186
- [Background] Lu KL, Chen S, Leung LP. Initial Experience of an Emergency Department in Shenzhen in Responding to the Emerging Wuhan Coronavirus Pneumonia. Ann Emerg Med. 2020 Apr;75(4):556. doi: 10.1016/j.annemergmed.2020.02.006. No abstract available. PMID 32216893
- [Background] Hu Y, Deng H, Huang L, Xia L, Zhou X. Analysis of Characteristics in Death Patients with COVID-19 Pneumonia without Underlying Diseases. Acad Radiol. 2020 May;27(5):752. doi: 10.1016/j.acra.2020.03.023. Epub 2020 Apr 7. No abstract available. PMID 32273135
- [Background] Chen C, Zhou Y, Wang DW. SARS-CoV-2: a potential novel etiology of fulminant myocarditis. Herz. 2020 May;45(3):230-232. doi: 10.1007/s00059-020-04909-z. No abstract available. PMID 32140732